CLINICAL TRIAL: NCT06974721
Title: Wearable Flexible Sensors for Spinal Motion Monitoring in Spinal Diseases
Brief Title: Wearable Flexible Sensors for Spinal Motion Monitoring
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: PekingUTH20250325
Record Dates: First submitted 2025-04-29; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-03

CONDITIONS: Spine Disease
Keywords: flexible sensor; spine disease
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
With the deepening of societal aging, degenerative spinal diseases have become increasingly prevalent in China and are one of the leading causes of disability among middle-aged and elderly populations. Current musculoskeletal assessment methods primarily focus on imaging rather than functional evaluation, and emphasize static over dynamic analysis, failing to capture the daily functional state of the musculoskeletal system. This limitation hinders a deeper understanding of functional patterns and their role in the progression of degenerative spinal diseases. Therefore, there is an urgent need to develop precise and dynamic functional assessment methods that overcome the constraints of time and space in measurement. This project adopts a dynamic perspective of the musculoskeletal system, developing a wearable monitoring approach based on flexible sensors to assess limb and spinal motion. The method will be validated against traditional imaging techniques such as X-ray and ultrasound, laying the foundation for investigating the pathogenesis of degenerative spinal diseases. This research aligns with China's strategic initiatives and practical needs in addressing the challenges of an aging population.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Spinal Cord Injury
2. Clinical diagnosis of cervical spondylotic myelopathy with Impaired Hand Function
3. Clinical diagnosis of Kyphosis
4. Clinical diagnosis of Spinal Imbalance
5. Clinical diagnosis of Scoliosis Patients
6. Clinical diagnosis of Lumbar Spondylolisthesis Patients

Exclusion Criteria:

1. Obesity (BMI>30)
2. Inability to complete functional assessments due to physical condition or other reasons;
3. Comorbid neuromuscular disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We are recruiting patients with spinal diseases, including cervical spondylosis with hand dysfunction, kyphosis/spinal imbalance, scoliosis (Cobb angle 20°-50°), and lumbar spondylolisthesis (>3mm dynamic slip).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Motor and Stabilizing Function of the Spine | Baseline
  The assessment of spinal stability at the baseline involves evaluating flexion-extension mobility in the sagittal plane, lateral bending capability in the coronal plane, and detecting relative displacement between vertebral segments during three-dimensional motion.

SECONDARY OUTCOMES:
Limb Motor Function | Baseline
  Assessment of Limb Muscle Strength Function Using Dynamometer Grip Strength Tests and Hand Function Scoring at the baseline.

REFERENCES:
- [Background] Wang Y, Zheng L, Yang J, Wang S. A Grip Strength Estimation Method Using a Novel Flexible Sensor under Different Wrist Angles. Sensors (Basel). 2022 Mar 4;22(5):2002. doi: 10.3390/s22052002. PMID 35271152
- [Background] Han G, Zhou S, Wang W, Li W, Qiu W, Li X, Fan X, Li W. Correlations between paraspinal extensor muscle endurance and clinical outcomes in preoperative LSS patients and clinical value of an endurance classification. J Orthop Translat. 2022 Sep 20;35:81-86. doi: 10.1016/j.jot.2022.08.005. eCollection 2022 Jul. PMID 36196076
- [Background] Li Z, Zhang S, Chen Y, Ling H, Zhao L, Luo G, Wang X, Hartel MC, Liu H, Xue Y, Haghniaz R, Lee K, Sun W, Kim H, Lee J, Zhao Y, Zhao Y, Emaminejad S, Ahadian S, Ashammakhi N, Dokmeci MR, Jiang Z, Khademhosseini A. Gelatin methacryloyl-based tactile sensors for medical wearables. Adv Funct Mater. 2020 Dec 1;30(49):2003601. doi: 10.1002/adfm.202003601. Epub 2020 Sep 6. PMID 34366759
- [Background] Hodges PW, Bailey JF, Fortin M, Battie MC. Paraspinal muscle imaging measurements for common spinal disorders: review and consensus-based recommendations from the ISSLS degenerative spinal phenotypes group. Eur Spine J. 2021 Dec;30(12):3428-3441. doi: 10.1007/s00586-021-06990-2. Epub 2021 Sep 20. PMID 34542672